CLINICAL TRIAL: NCT02908217
Title: Safety and Efficacy of tocilizuMAb Versus Placebo in Polymyalgia rHeumatica With glucocORticoid dEpendence SEMAPHORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Roche Chugai (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SEMAPHORE (RB15.210)
Record Dates: First submitted 2016-09-16; First posted 2016-09-20 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Polymyalgia Rheumatica
Keywords: Polymyalgia Rheumatica; Tocilizumab; Glucocorticoid
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (Experimental): 6 Intravenous infusions of tocilizumab in a dosage of 8 mg/kg (or 4 mg/kg depending on biological results as mentioned by the SPC of Tocilizumab for the rheumatoid arthritis) every 4 weeks.
  Interventions: Drug: Tocilizumab
- Placebo (Placebo Comparator): 6 Intravenous infusions of placebo (sterile sodium chloride solution) every 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tocilizumab — 6 Intravenous infusions of tocilizumab in a dosage of 8 mg/kg (or 4 mg/kg depending on biological results as mentioned by the SPC of Tocilizumab for the rheumatoid arthritis) every 4 weeks.
  Other Names: Intravenous infusions of tocilizumab
  Arms: Tocilizumab
Drug: Placebo — 6 Intravenous infusions of placebo every 4 weeks.
  Other Names: Intravenous infusions of placebo
  Arms: Placebo

SUMMARY:
Patients are treated with infusions of Tocilizumab (TCZ) or placebo for 5 months. Clinical evaluation is performed using PMR-AS.

The PMR-AS is computed by summing the 5 variables after multiplying by 0.1 for weighting purposes: PMR-AS (activity scale = AS) = C reactive protein (CRP) (mg/dl) + patient scale (VASp) (0-10 scale) + physician scale (VASph) (0-10 scale) + morning stiffness(MST) [min]×0.1) + elevation of upper limbs (EUL) (0-3 scale).

All the patients included are treated with glucocorticoid (GC).GC are reduced at each visit until the end of the study, depending on response to treatment and PMR-AS.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 50 years
* Fulfilled the Chuang criteria
* And currently:

  * PMR-AS> 10
  * Absence of signs or symptoms of other musculoskeletal or connective tissue conditions
* Able to give informed consent
* Concomitant treatments with methotrexate or hydroxy-chloroquine are permitted if stable dose since 3 months.

Exclusion Criteria:

* Clinical symptoms of giant cell arteritis
* Uncontrolled dyslipidemia, high blood pressure or cardiovascular disease
* History of major organ or haematopoietic stem cell/marrow transplant
* Clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to PMR
* Planned surgical procedure within 12 months after randomization.
* History of malignant neoplasm within the last 5 years.
* Current active infection
* Patient with elevated ALT or AST> 5 ULN

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Low disease activity (PMR-AS<10) with steroid independence (GCs ≤5 mg absolute value) or decrease ≥ 10 mg from week 0 to week 24). | From week 0 to week 24
  PMR-AS measure

SECONDARY OUTCOMES:
Proportion of patients with (PMR-AS>17) in both arm | From Week 24 to Week 32
  PMR-AS measure
PMR-AS and proportion of patients with PMR-AS < 1.5; 10; 17. | From inclusion to week 32
  PMR-AS measure
Cumulative dosages of GCs at Week 32 | Week 32
  dosages of GCs

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Devauchelle-Pensec, Pr, Principal Investigator — CHRU de Brest
Locations (17):
- France (17):
  - Hopital Nord service de rhumatologie-Franche Comté, Belfort
  - CIC Besançon, Besançon
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHRU Brest, Brest
  - Centre hospitalier Sud-Francilien, Corbeil-Essonnes
  - CHU Dijon, Dijon
  - CH Le Mans, Le Mans
  - Hôpital européen, Marseille
  - Ch Des Pays de Morlaix, Morlaix
  - CH Mulhouse, Mulhouse
  - CHU de Nancy, Nancy
  - CHU Nantes, Nantes
  - hôpital Sapêtrière -APHP, Paris
  - CHU Rennes, Rennes
  - CHU St Etienne, Saint-Etienne
  - CHRU de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Devauchelle-Pensec V, Carvajal-Alegria G, Dernis E, Richez C, Truchetet ME, Wendling D, Toussirot E, Perdriger A, Gottenberg JE, Felten R, Fautrel BJ, Chiche L, Hilliquin P, Le Henaff C, Dervieux B, Direz G, Chary-Valckenaere I, Cornec D, Guellec D, Marhadour T, Nowak E, Saraux A. Effect of Tocilizumab on Disease Activity in Patients With Active Polymyalgia Rheumatica Receiving Glucocorticoid Therapy: A Randomized Clinical Trial. JAMA. 2022 Sep 20;328(11):1053-1062. doi: 10.1001/jama.2022.15459. PMID 36125471